CLINICAL TRIAL: NCT01751958
Title: Phase 3 Study of Evaluate Radiation Exposure and Procedure Times for Continuous Fluoroscopic Monitoring During Lumbar ESI
Brief Title: Radiation Exposure in Spine Intervention Under Angiography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Suyoung Kim, Researcher, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1105/128-014
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural Steroid injection (Experimental): Group-Epidural Steroid injection (Intermittent)
  Interventions: Radiation: Epidural steroid injection
- Epidural Steroid Injection2 (Experimental): Group-injection under angiography (continuous)
  Interventions: Radiation: Epidural steroid injection

INTERVENTIONS:
Radiation: Epidural steroid injection — Epidural steroid injection

SUMMARY:
Evaluate radiation exposure and procedure times for continuous fluoroscopic monitoring during lumbar ESI

DETAILED DESCRIPTION:
The purpose of this prospective study was to evaluate radiation exposure and procedure times for fluoroscopic monitoring during lumbar ESI with analyzing the differences among operators (experienced staff and trainee) and among different method for ESI.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of having radiculopathic low back pain

Exclusion Criteria:

* Angiography is contraindicated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Radiation dose | Treatment on the day
  Radiation dose of patients with spine invervention under angiography

CONTACTS AND LOCATIONS:
Overall Officials: Joon-woo Lee, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Joon-woo Lee, Seongnam-si, Gyeonggi-do, South Korea